CLINICAL TRIAL: NCT00186186
Title: Depakote ER in Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Abbott (Industry); National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Terrence Ketter, Professot, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 79130
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Depression, Bipolar
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Depakote ER (Experimental): Depakote ER up to 1500 mg/day
  Interventions: Drug: Depakote ER

INTERVENTIONS:
Drug: Depakote ER — Depakote ER

SUMMARY:
The purpose of this study is to examine the safety and efficacy of Depakote ER in bipolar depression and to evaluate metabolic and GABA changes with Depakote ER administration using PET and MRI/MRS brain imaging techniques.

DETAILED DESCRIPTION:
Mood disorders are important public health problems. Bipolar disorder is a major psychiatric disorder characterized by mood cycles alternating between mania and depression and affects approximately 1% of the population. Most patients are treated beginning in the early twenties and then embark on a course marked by multiple recurrences, hospitalizations, and encounters with legal authorities. These disorders inflict substantial morbidity which yields important deficits in occupational and interpersonal function. The risk of suicide in mood disorders may be as high as 10%.

Although the outlook for recovery from acute manic or depressive episodes is generally excellent, the long-term prognosis of the disorder varies tremendously across the patient population. The introduction of lithium, anticonvulsants and atypical antipsychotics significantly changes the outlook for bipolar disorder, with some individuals on chronic treatment attaining complete remission and indefinite prophylaxis against mood episodes. However, such optimum outcomes may be limited to as few as one-third to one-half of all treated patients. The remaining experiences various combinations of breakthrough mood episodes, including chronic mood instability, persistent depression, and rapid cycling.

Very little research has been conducted with bipolar disorder, and no medications have an FDA indication to treat bipolar depression. Previous studies suggest that Depakote is promising in the treatment of mixed and depressed episodes of bipolar disorder. This study utilizes the extended release formulation of divalproex sodium, with demonstrated increased tolerability.

We propose investigating safety, tolerability and efficacy of Depakote ER monotherapy in Bipolar I, II or NOS depression, and monitoring associated changes in brain GABA levels. In addition, we intend to evaluate and assess the differences between brain metabolic rate and GABA levels in bipolar disorder patients and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I, II or NOS currently suffering from depression
* Both: both female and male participants are being studied
* Adults 18 years and older of any race

Exclusion Criteria:

* Schizophrenia or schizoaffective disorder and other disorders excluded at the discretion of the investigator's discretion
* Substance dependence within the past 3 months and abuse within the past 2 weeks prior to study.
* Positive screen for psychoactive drugs, stimulants or drugs of abuse (excluding marijuana, as long as dependence and abuse are ruled out according to DSM-IV)
* Significant risk harm to self or others based on history and mental status exam
* Clinically significant or unstable medical condition
* Unstable thyroid pathology and treatment initiated or altered within the past 3 months
* Clinically significant abnormal laboratory test results, vital signs, as judged by the investigators
* Women pregnant or nursing, or WOCBP who do not use adequate contraception or who are judged to be unreliable in their use of contraception
* Subjects who failed (because of inefficacy or adverse effects) an adequate trial of Depakote; eligible patient's may not have received Depakote within 30 days of screen

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence A. Ketter, MD, Study Director — Stanford University, Department of Psychiatry and Behavioral Sciences
Locations (1):
- Stanford University Bipolar Disorders Clinic, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang PW, Nowakowska C, Chandler RA, Hill SJ, Nam JY, Culver JL, Keller KL, Ketter TA. Divalproex extended-release in acute bipolar II depression. J Affect Disord. 2010 Jul;124(1-2):170-3. doi: 10.1016/j.jad.2009.10.021. PMID 19923006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were recruited from the Bipolar Disorders Clinic at the Stanford University School of Medicine in Stanford, California. Patients met DSM-IV criteria for bipolar II disorder, with a current major depressive episode, as determined by the Systematic Treatment Enhancement for Bipolar Disorder (STEP-BD)
Groups:
- Depakote ER: Open-label. All subjects received Depakote extended release (ER) starting 250mg/daily at bedtime. Dose was increased every 4 days by 250mg/day as necessary and tolerated up to 1500 mg/day. All subjects took medication over a period of 7 weeks or terminated at the final visit (whichever came first).
Period: Overall Study
Arm/Group | Depakote ER
Started | 28
Completed | 20
Not Completed | 8
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 3
Not completed — Not reported as to reason | 2

BASELINE CHARACTERISTICS:
Arm/Group | Depakote ER
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 28
Montgomery Asberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders.
  Higher MADRS score indicates more severe depression the overall score ranges from 0 to 60.
  Usual cutoff points are:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression.
  units on a scale | 30.1 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders.
  Higher MADRS score indicates more severe depression the overall score ranges from 0 to 60.
  Usual cutoff points are:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression.
Time Frame: Baseline, 7 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depakote ER
Number analyzed (Participants) | 20
units on a scale | 14.9 (9.8)
Statistical Analysis 1: Comparison: Depakote ER; Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Response to the Divalproex-ER in Acute Bipolar 2 Depression.
Description: A reduction greater than or equal to 50% in MADRS total score from baseline to the endpoint.
Time Frame: 7 weeks
Measure: Number; unit: participants
Arm/Group | Depakote ER
Number analyzed (Participants) | 20
participants | 11
Statistical Analysis 1: Comparison: Depakote ER; Test type: Superiority or Other; Percentage = 54

ADVERSE EVENTS:
Arm/Group | Depakote ER
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 3/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Depakote ER (N=28)
Weight gain (Metabolism and nutrition disorders) | 3 (3) — ≥ 7% Weight gain

LIMITATIONS AND CAVEATS:
This trial is limited by small sample size, as well as an open-label study design with no placebo control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No